CLINICAL TRIAL: NCT04416204
Title: Role of Hepatic Glycogen on Nocturnal EGP in T2D
Brief Title: Effect of High Carbohydrate vs. Low Carbohydrate Diet in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Mayo Clinic (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rita Basu, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 22074; R01DK029953 (NIH)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; hepatic glycogen; endogenous glucose production
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Masking Description: A total of 34 subjects participated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 diabetes (Experimental): Participants with Type 2 Diabetes received Glycogen loading (GL) and Non-Glycogen loading (NGL) meal in a randomized manner.
  Interventions: Other: glycogen loading; Other: No Glycogen Loading
- Participants without diabetes (Experimental): Participants with no Diabetes received Glycogen loading (GL) and Non-Glycogen loading (NGL) meal in a randomized manner.
  Interventions: Other: glycogen loading; Other: No Glycogen Loading

INTERVENTIONS:
Other: glycogen loading — Subjects will consume an isocaloric diet [60% carbs, 20% protein, 20% fat (33 kcal/kg/day)] for 3 days prior to the overnight study.
Other: No Glycogen Loading — Subjects will consume an isocaloric diet [40% carbs, 20% protein, 40% fat (33 kcal/kg/day)] for 3 days prior to the overnight study.

SUMMARY:
The experimental approach in this study intends to investigate the role of hepatic glycogen content on nocturnal regulation of endogenous glucose production including the relative contributions of glycogenolysis and gluconeogenesis and the extent to which this differs between subjects with type 2 diabetes and subjects without diabetes. Both participants with type 2 diabetes and participants without diabetes will be studied after consuming either a low carbohydrate (no glycogen loading) or high carbohydrate (glycogen loading) diet.

DETAILED DESCRIPTION:
Physiology study for looking at glycogen loading vs non loading in improving nightime glucose tolerance by increasing glycogen in liver and resulting higher glycogenolysis at night.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-75
* BMI 20-35kg/m^2
* Participants with type 2 diabetes:

  * HbA1c less than or equal to 8.5% on lifestyle therapy or monotherapy with metformin or sulphonylureas (SU); or less than or equal to 7.5% on two oral hypoglycemic agents (Metformin and SU)

Exclusion Criteria:

* Pregnancy or breast feeding
* Morbidities precluding participation
* Participants with type 2 diabetes:

  * Therapy with insulin
  * SGLT2 inhibitors
  * GLP-1 based approaches
  * TZDs
  * Unstable diabetic retinopathy
  * Microalbuminuria
  * Macrovascular disease
  * Medications affecting GI motility (eg., erythromycin, pramlintide)
  * Upper GI disorder/surgery
* Participants without diabetes:

  * Medications (except stable thyroid hormone or hormone replacement therapy) that could influence glucose tolerance
  * History of diabetes mellitus in first degree family members or prior history of diabetes mellitus or gestational diabetes, or pre-diabetes

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 Type 2 Diabetes subjects were screened, 1 subject did not meet eligibility criteria, 2 subjects withdrew from the study.
  17 subjects without Diabetes were screened, 2 subjects withdrew from the study.
Pre-assignment Details: Subject enrolled after consent were screened to meet inclusion criteria. If not met subjects were excluded.
  14 Type 2 Diabetes and 15 without Diabetes subjects were randomized to receive, either Glycogen loading or Non-Glycogen loading meal during visit 1. All subjects were tested for Glycogen loading and Non-Glycogen loading meal in a randomized order.
  1Type 2 Diabetes and 2 without Diabetes subjects did not participate in visit 2.
Groups:
- Type 2 Diabetes - GL Then NGL: Participants with Type 2 Diabetes received Glycogen loading (GL) followed by Non-Glycogen loading (NGL) meal after 3-6 weeks of washout
- Type 2 Diabetes - NGL Then GL: Participants with Type 2 Diabetes received Non-Glycogen loading (NGL) followed by Glycogen loading (GL) meal after 3-6 weeks of washout
- Participants Without Diabetes - GL Then NGL: Participants with no Diabetes received Glycogen loading (GL) followed by Non-Glycogen loading (NGL) meal after 3-6 weeks of washout
- Participants Without Diabetes - NGL Then GL: Participants with no Diabetes received Non-Glycogen loading (NGL)followed by Glycogen loading (GL) meal after 3-6 weeks of washout
Period: First Visit
Arm/Group | Type 2 Diabetes - GL Then NGL | Type 2 Diabetes - NGL Then GL | Participants Without Diabetes - GL Then NGL | Participants Without Diabetes - NGL Then GL
Started | 6 | 8 | 7 | 8
Completed | 6 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Washout (3-6 Weeks)
Arm/Group | Type 2 Diabetes - GL Then NGL | Type 2 Diabetes - NGL Then GL | Participants Without Diabetes - GL Then NGL | Participants Without Diabetes - NGL Then GL
Started | 6 | 8 | 7 | 8
Completed | 5 | 8 | 6 | 7
Not Completed | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Period: Second Visit
Arm/Group | Type 2 Diabetes - GL Then NGL | Type 2 Diabetes - NGL Then GL | Participants Without Diabetes - GL Then NGL | Participants Without Diabetes - NGL Then GL
Started | 5 | 8 | 6 | 7
Completed | 5 | 8 | 6 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Type 2 Diabetes: High Carbohydrate (glycogen loading): Subjects will consume an isocaloric diet [60% carbs, 20% protein, 20% fat (33 kcal/kg/day)] for 3 days prior to the overnight study.
  Low carbohydrate (No Glycogen Loading): Subjects will consume an isocaloric diet [40% carbs, 20% protein, 40% fat (33 kcal/kg/day)] for 3 days prior to the overnight study.
  Baseline characteristics of all subjects with Type 2 Diabetes reported.
- Participants Without Diabetes: High Carbohydrate (glycogen loading): Subjects will consume an isocaloric diet [60% carbs, 20% protein, 20% fat (33 kcal/kg/day)] for 3 days prior to the overnight study.
  Low carbohydrate (No Glycogen Loading): Subjects will consume an isocaloric diet [40% carbs, 20% protein, 40% fat (33 kcal/kg/day)] for 3 days prior to the overnight study.
  Baseline characteristics of all subjects without Diabetes reported.
- Total: Total of all reporting groups
Arm/Group | Type 2 Diabetes | Participants Without Diabetes | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (7.7) | 54.5 (14.0) | 58.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Weight (Kg) [Mean (Standard Deviation); unit: Kg] | 82.4 (11.0) | 82.5 (12.5) | 82.4 (11.6)
BMI (Kg/m^2) [Mean (Standard Deviation); unit: Kg/m^2] | 28.0 (2.8) | 28.5 (2.9) | 28.2 (2.8)
Fasting Plasma Glucose (mmol/L) [Mean (Standard Deviation); unit: mmol/L] | 8.0 (3.5) | 4.7 (0.4) | 6.3 (2.9)
HbA1C [Mean (Standard Deviation); unit: % of Glycosylated Haemoglobin] | 7.1 (1.4) | 5.3 (0.4) | 6.2 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Glycogen Content and Rates of Gluconeogenesis in Subjects With Type 2 Diabetes
Description: We measured the rates and contribution of Gluconeogenesis (GNG) to nocturnal Endogenous Glucose Production (EGP) using the deuterated water technique after either glycogen loading or no glycogen loading in subjects with type 2 diabetes.
Time Frame: Subjects will complete both glycogen loading and no glycogen loading visits within approximately 6 weeks
Population: Gluconeogenesis (GNG) and Endogenous Glucose Production (EGP) measured after glycogen loading (GL) or no glycogen loading (NGL) in subjects with type 2 diabetes.
Measure: Mean (Full Range); unit: umol/kgFFM/min
Groups:
- Type 2 Diabetes - Glycogen Loading: Type 2 Diabetes after a Glycogen Loading meal
- Type 2 Diabetes - Non-Glycogen Loading: Type 2 Diabetes after a Non-Glycogen Loading meal
Arm/Group | Type 2 Diabetes - Glycogen Loading | Type 2 Diabetes - Non-Glycogen Loading
Number analyzed (Participants) | 14 | 13
umol/kgFFM/min
  GNG (umol/kgFFM/min) | 8.2 [7.0 to 9.4] | 9.4 [8.2 to 10.5]
  EGP (umol/kgFFM/min) | 17.4 [16.0 to 18.7] | 15.6 [14.2 to 17.0]

2. Secondary Outcome: Rates of Glycogenolysis in Subjects With Type 2 Diabetes
Description: Rates and contribution of glycogenolysis (GLY) to nocturnal EGP will be measured using the deuterated water technique after glycogen loading and no glycogen loading in subjects with type 2 diabetes.
Time Frame: Subjects will complete both glycogen loading and no glycogen loading visits within approximately 6 weeks
Population: Glycogenolysis (GGL) and Endogenous Glucose Production (EGP) measured after glycogen loading (GL) or no glycogen loading (NGL) in subjects with type 2 diabetes.
Measure: Mean (Full Range); unit: umol/kgFFM/min
Arm/Group | Type 2 Diabetes - Glycogen Loading | Type 2 Diabetes - Non-Glycogen Loading
Number analyzed (Participants) | 14 | 13
umol/kgFFM/min
  GGL (umol/kgFFM/min) | 9.2 [7.6 to 10.8] | 6.3 [4.7 to 7.9]
  EGP (umol/kgFFM/min) | 17.4 [16.0 to 18.7] | 15.6 [14.2 to 17.0]

3. Secondary Outcome: Rates of Gluconeogenesis in Healthy Subjects
Description: Rates of GNG will be measured through the night using the deuterated water technique after either glycogen loading or no glycogen loading in healthy subjects.
Time Frame: Subjects will complete both glycogen loading and no glycogen loading visits within approximately 6 weeks
Population: Gluconeogenesis (GNG) and Endogenous Glucose Production (EGP) measured after glycogen loading (GL) or no glycogen loading (NGL) in subjects without diabetes.
Measure: Mean (Full Range); unit: umol/kgFFM/min
Groups:
- Participants Without Diabetes - Glycogen Loading: Participants without Diabetes after a Glycogen Loading meal
- Participants Without Diabetes - Non- Glycogen Loading: Participants without Diabetes after a Non- Glycogen Loading meal
Arm/Group | Participants Without Diabetes - Glycogen Loading | Participants Without Diabetes - Non- Glycogen Loading
Number analyzed (Participants) | 13 | 14
umol/kgFFM/min
  GNG (umol/kgFFM/min) | 7.7 [6.5 to 8.9] | 8.5 [7.3 to 9.7]
  EGP(umol/kgFFM/min) | 15.9 [14.5 to 17.2] | 13.5 [12.1 to 14.8]

ADVERSE EVENTS:
Time Frame: Across the study duration. GL or NGL meal for a period of 3 days and an overnight infusion protocol, followed by washout for approximately 3-6 weeks. Second visit GL or NGL meal for a period of 3 days and an overnight infusion protocol.
Description: There are no safety endpoints as there were no drugs involved and study risks were limited to that of blood draw only.
Groups:
- Participants Without Diabetes - NGL Then GL: Participants with Type 2 Diabetes received Non-Glycogen loading (NGL) followed by Glycogen loading (GL) meal after 3-6 weeks of washout
Arm/Group | Type 2 Diabetes - GL Then NGL | Type 2 Diabetes - NGL Then GL | Participants Without Diabetes - GL Then NGL | Participants Without Diabetes - NGL Then GL
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/7 | 0/8

LIMITATIONS AND CAVEATS:
• Though unlikely, it is possible that additional steps to load hepatic glycogen maybe necessary (e.g., late night snack: high carb in GL and isocaloric low carb in NGL) to maximize differences in liver glycogen contents between visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT04416204/Prot_SAP_000.pdf